CLINICAL TRIAL: NCT05420103
Title: Research Proposal of New Technologies and Standardization of Physiotherapy Stroke Rehabilitation - A Retrospective Functional Outcomes Analysis of Accelerated Stroke Ambulation Program (ASAP)
Brief Title: Research Proposal of New Technologies and Standardization of Physiotherapy Stroke Rehabilitation
Status: Completed | Type: Observational
Sponsor: Tai Po Hospital (Other Government)
Responsible Party: Principal Investigator, Bryan Ping Ho CHUNG, Senior Physiotherapy, Tai Po Hospital
Other Study IDs: NTEC-2022-0267
Record Dates: First submitted 2022-06-08; First posted 2022-06-15 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Stroke
Keywords: stroke; rehabilitation; physiotherapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-ASAP: Conventional Stroke Rehabilitation Program
- Post-ASAP: Standardized functional assessment, standardized intensive early ambulation with modern technologies such as Knee-Ankle-Foot Orthoses and Robotic-Assisted Gait Training. In order to monitor the progress of each patient proactively, Stroke Registry and Reference Modified Rivermead Mobility Index (MRMI) Gain were developed. Stroke Registry was a longitudinal stroke rehabilitation database to monitor patients' functional outcomes and therapists' intervention compliance so as to pave the way for future clinical big data movement to bridge the gap between evidence-practice and clinical practice. Reference MRMI Gain was a clinical prediction model apply business intelligence concept to support goal-orientated approach of physiotherapists in stroke rehabilitation. Stroke treatment library, a standardized exercise prescription in video format was also developed to facilitate standardized prescription of interventions to patients with different level of ability.
  Interventions: Other: Accelerated Stroke Ambulation Program

INTERVENTIONS:
Other: Accelerated Stroke Ambulation Program — Stroke Rehabilitation Program
  Groups: Post-ASAP

SUMMARY:
One of the main goals of physiotherapy in stroke rehabilitation is to maximize walking ability of patients as soon as possible. Traditionally, intervention selection and application of neuroplasticity to stroke patients depends on personal preference and experience of therapists. Recent development of technologies may provide more accessible, efficient, objective, intensive and predictive methods compared to traditional practices in facilitating the process of recovery after brain injury and standardizing stroke rehabilitation programs.

A clinical quality improvement program named Accelerated Stroke Ambulation Program (ASAP) was started in Stroke Rehabilitation Program Tai Po Hospital by Physiotherapy Department since 2019, pilot period from October 2019 to September 2020 and execute as standard practice afterward.

DETAILED DESCRIPTION:
The goal of ASAP was to facilitate maximal walking ability of stroke patients by standardized application of modern technologies. ASAP features standardized functional assessment, standardized intensive early ambulation with modern technologies such as Knee-Ankle-Foot Orthoses, Lower Limb Robotic-Assisted Gait Training and Video-Guide Training. In order to monitor the progress of each patient proactively, Stroke Registry and Reference Modified Rivermead Mobility Index (MRMI) Gain were developed. Stroke Registry was a longitudinal stroke rehabilitation database to monitor patients' functional outcome and therapists' intervention compliance. Reference MRMI Gain was a clinical prediction model based on big data concept to support goal-orientated approach of physiotherapists in stroke rehabilitation. Stroke treatment library, a standardized exercise prescription in video format was also developed to facilitate standardized prescription of interventions to patients with different level of ability.

ELIGIBILITY:
Inclusion Criteria:

Patients with principal diagnosis of cerebrovascular accident, stroke, or hemiplegia and had received has received physiotherapy gym session training in a hospital in Hong Kong between the periods from 1 October 2018 to 31 September 2019 and from 1 October 2020 to 31 September 2021.

Exclusion Criteria:

Transfer out of the hospital, discharged against medical advice or died.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with principal diagnosis of cerebrovascular accident, stroke, or hemiplegia and had received has received physiotherapy gym session training in a hospital in Hong Kong between the periods from 1 October 2018 to 31 September 2019 and from 1 October 2020 to 31 September 2021.
Sampling Method: Non-Probability Sample
Enrollment: 650 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2022-06-08 (Actual)

PRIMARY OUTCOMES:
Modified Rivermead Mobility Index | The first day of assessment
  Modified Rivermead Mobility Index consists of eight test items, including turning over, changing from lying to sitting, maintaining sitting balance, going from sitting to standing, standing, transferring, walking indoors, and climbing stairs. The score of MRMI range from 0 to 40, the higher score the more independence in mobility.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Ping Ho CHUNG, Principal Investigator — Tai Po Hospital
Locations (1):
- Tai Po Hospital, Hong Kong, Hong Kong